## Vietnam Cryptococcal Retention in Care Study (CRICS)

## **CASE REPORT FORMS**

Ver 2.1

### **Identifying information:**

FOA No: GH-12-008

Award Number: GH 000758

Date: 7 January, 2017

### **APPENDIX 1: SCREENING FORM (Phase 1 only)**

| Patient's name: | Patient's name:Male/Female: |
|---|---|
| Date and selection criteria | |
| Screening date | / / (dd/mm/vv) |
| Age of patient | |
| History of ART treatment | <ul> <li>&lt;18 years old → Patient does not meet the selection</li> <li>Have never taken ARVs</li> <li>Has taken ARVs in the past, but has not had &gt;4 consecutive weeks of ARVs in the past year.</li> <li>Has been taking ARVs for more than 4 consecutive weeks in the past 1 year → Patient does not meet the</li> </ul> |
| History of prior / current CM (or current treatment for CM) | <ul><li>No</li><li>Yes → Patient does not meet the selection criteria</li></ul> |
| Receipt of systemic antifungal medication for more than 4 consecutive weeks within the past 6 months | <ul><li>No</li><li>Yes → Patient does not meet the selection criteria</li></ul> |
| For woman patient: Are you currently pregnant or planning to become pregnant during the next 2 years? | <ul><li>No</li><li>Yes →If CrAg positive, patient is not eligible to participate in the study.</li></ul> |
| INFORMATION FOR PATIENTS | |
| What is cryptococcal disease?: A fungal is especially in people living with HIV - Are you HIV positive and 18 years old - Today your CD4 is less than or equal | |
| If you are HIV-positive, are at least 18 years old, and your CD4 is less than or equal to 100 cells/ $\mu$ L, the Vietnam Ministry of Health and the World Health Organization recommend that your blood should be screened for "Crypto," a fungal disease that can affect the brain. | |
| second time to take another sample if yo | CD4 testing. To save time and to avoid your coming back a ur CD4 is $\leq 100$ cells/ $\mu$ L, we will use a small amount of the er laboratory tests to check if you have "Crypto". |
| For more information, please ask your nu | rse or clinician during this visit. |

#### APPENDIX 2A: SCRIPT FOR INFORMING PATIENTS ABOUT CRAG SCREENING

There is an organism called Cryptococcus, or "Crypto" for short that can cause disease in people and can affect the brain, lungs, and other parts of the body. People are more likely to get Crypto if they have HIV and low immunity, i.e., CD4 counts, less than 100 cells/µL. For those who have Crypto, at the early infection stage, they may not have any clinical symptoms (called asymptomatic patients) but lately when symptom appear, they will become seriously ill. In order to prevent people from getting ill with Crypto brain and lung infections, we are testing patients who have low CD4 counts to determine if they may already have the fungus in blood. This will allow us to treat early and prevent serious illness. If the test shows that you have early Crypto, we will contact you as soon as we can to assess whether to start you on treatment.

- a. "We will perform routine screening for Crypto on all patients with CD4 counts, less than 100 cells/ $\mu$ L and we'll be doing that from the blood that remains after CD4 testing.
- b. If you have already had a CD4 test done within the last 2 weeks, the leftover plasma from other routine tests collected today will be used.
- c. If no other tests are requested today, a small blood sample will be taken for CrAg screening."
- d. "You will be informed of your CrAg results at the same time as your CD4 results or a separate CrAg result if you already had CD4 counts previously tested less than or equal to 100 cells/μL"
- e. "If your CrAg test is positive, we will provide treatment to prevent you from developing severe disease unless your doctors think that you may be harmed due to the treatment."

Do you have any questions?

#### APPENDIX 3A: INFORMED CONSENT FORM

#### **PART I: Information Sheet**

#### Introduction

Hello. My name is (name of study officer) . I would like to talk to you about a research study we are doing and to ask if you would want to take part in it. This study is sponsored by the United States Centers for Disease Control and Prevention (CDC). The investigators, who are doctors at National Hospital for Tropical Diseases and Tropical Diseases Hospital, will be responsible for the study. Hundreds of patients are expected to be included in the study at over 22 sites throughout Vietnam. If you do not understand something, please ask me to stop and to tell you again or to answer any questions you may have.

#### Purpose of the research

There is an organism called Cryptococcus, or "Crypto" for short, which can cause fungal disease in people, especially people with HIV. The disease can affect the brain and the breathing system. We are doing a study of people with HIV, to see if certain new ways of testing for and treating early Crypto infection with a medicine called fluconazole can help prevent patients from getting very sick. The information we learn will be used to try to help other people with HIV.

#### **Participant selection**

We are asking many patients with HIV infection if they would like to take part in this study. You are invited to take part in the study because you:

- Are aged  $\geq$  18 years,
- Are a patient at one of the HIV clinics in Vietnam taking part in the study
- Have advanced HIV disease (as shown by having a CD4 count less than 100 cell/μL)
- Are about to start taking medicine called ART for HIV infection

Pregnant women cannot take fluconazole because fluconazole can damage a developing fetus. If you are female, and you test positive for Crypto, you will be required to have a pregnancy test before you begin this study treatment; if it turns out that you are pregnant or if you plan to become pregnant in the next 2 years you cannot be in the study if you have crypto in your blood. If you are sexually active, we encourage you to use a modern contraceptive method, such as the contraceptive pill, during the course of the study to avoid becoming pregnant while on fluconazole.

#### **Voluntary Participation**

Taking part in this study is your choice. If you do not to take part in the study, you will receive the same care that all patients here usually get. If you decide to be in the study, you may change your mind later and stop being in the study. If you decide to stop taking part, you will receive the same care that all patients here usually get.

#### **Study Procedures**

This study will be conducted as part of routine procedures at the clinic. In addition to the information doctors will ask in order to provide care, some additional information will be required during the study. Answering these questions may take an additional 20-30 minutes each visit. For the study, we will follow you for at least 6 months and up to 12 months after ART initiation and at we will collect some additional information from you at these visits. If you test positive for Crypto, you will be asked to come to the study clinic at the time you are enrolled (baseline), at 2 weeks, 10 weeks after study enrolment, and2 months, 6 months, and 12 months after ART initiation. If you test negative for CrAg, you will be asked to come to the study clinic at the time you are enrolled (baseline), at 2 months, 6 months, and 12 months after your ART initiation.

If you have a positive blood test for Crypto: This means you have a Crypto infection in the blood and are at higher risk for developing a Crypto brain infection. We will ask you some questions to see if you might have a Crypto brain infection right now. If you do, your doctor will be responsible for determining the best management of your disease according to national guidelines in Viet Nam.

If you do not have a Crypto brain infection, you still need medicine to help keep you from getting a Crypto brain infection. As part of this study, you will be given a drug called fluconazole to fight Crypto. You take this drug by mouth. First you will take 900 mg each day for 2 weeks, then450 mg each day for 8 weeks. After that, you will take 200 mg for 6 months and then 150 mg each day until your doctor lets you know it is safe to stop. This will be when you're immune system is strong enough to fight Crypto on its own.

If you have a negative blood test for Crypto: this means you probably do not have a Crypto infection at the moment. But, you might still get Crypto in the future if your immune system stays weak. Coming to the clinic for your appointments will let doctors check you for symptoms of Crypto and other diseases that people with HIV sometimes get.

#### **General Information**

If you are in this study, someone on the study team will look at your clinic medical chart to find out more about your health. Also, we will ask you some questions about yourself and your health before you came to the clinic. We will ask if you have been sick and why you came to the clinic. We will also look at your lab test records and, if you go to a hospital, your chart in the hospital. You can refuse to answer any questions you want and this will not affect the care you will get. If you become ill during this study and your doctor thinks that you might have a Crypto brain infection, your doctor will be responsible for determining the best management of your infection in accordance with Viet Nam national guidelines.

#### **Duration**

You will come to the clinic for regular visits like all HIV patients here. At the end of 12 months, the study will be done. While the study is going on, if you are in hospital and cannot come to the clinic for an appointment, please let us know. I would like to be able to contact you, or someone who lives with you, during the year that you are in the study, to remind you about your appointments for your clinic visits.

#### **Risks**

Fluconazole is a medicine that is used around the world to treat fungal infections, including Crypto. People taking fluconazole generally feel fine, but they might sometimes have an upset stomach, loose stools, headache, or a skin rash.

High doses of fluconazole, as used in this study, should not be used during the first three months of pregnancy because it can harm an unborn baby. If you think you have become pregnant while using this medicine, stop fluconazole immediately and tell your doctor right away. For women receiving fluconazole, at each follow up visit, your doctor will ask you about your last normal menstrual period (LNMP) and contraceptive use. If your LNMP is more than 5 weeks, you will be asked to undergo a pregnancy test. If the test is positive, your treatment with fluconazole will be stopped.

For patients who have liver disease, fluconazole can damage the liver. Signs that the liver is damaged include stomach pain on the right side, nausea or vomiting, and a yellow color of the skin and eyes. Please let the study doctors know if you or a friend or family member thinks your skin color has changed or if you have stomach pain, nausea, or vomiting. If you take fluconazole, the study team will watch carefully for possible side effects of the drug at each study visit.

If you get sick or have concerns or questions between your regular visits to clinic, please let us know by coming to the clinic for a check-up.

#### **Benefits**

If your test shows that you have Crypto infection, but you do not have symptoms, you will get medicine to treat Crypto for free. If you do have symptoms, your doctor will be responsible for determining the best management of your disease in accordance with Vietnam national guidelines. We will also use the information from you and many other patients to try to improve the health of all people living with HIV.

#### Reimbursements

We will give you 65000 Vietnam Dong [approximately US\$3]to pay for your extra time spent with us to answer questions regarding your quality of life for the study in your visit at 0, 6, and 12 months after your enrolment.

#### **Confidentiality**

Only your health care providers and the study team will know the information we collect or that you are in the study. We will not share your name or information about you with anyone else. If information is shared with other people who do not work with the study, your name will not be used and no one would be able to identify you.

#### Right to Refuse or Withdraw

You do not have to be in this study. If you do not want to be in this study, you can still come to this clinic and you will still get the regular care. You may stop being in the study at any time and you will not lose your rights as a patient here. Your treatment at this clinic will not be affected in any way.

#### Who to Contact

If you have questions, you may ask them now or later, even after the study has started. If you want to ask questions later, you can come to the clinic or you can contact any of the following: [name, address/telephone number/e-mail].

This protocol has been reviewed and approved by the Institutional Review Board (IRB) of the National Hospital for Tropical Diseases, the Tropical Diseases Hospital in Ho Chi Minh City, and the US Centers for Disease Control and Prevention in Atlanta, Georgia. This is a committee whose job is to protect people and make sure that they are not harmed in a study. If you wish to find about more about the IRB, contact National Hospital for Tropical Diseases at 78 Giai Phong street – Dong Da district, Hanoi, Vietnam, Tel: (84-4).35763491

You can ask me any more questions about any part of this research study, if you wish to. Do you have any questions?

#### **PART II: Consent Statement**

I have read the information about this study or it has been read to me. I have had the chance to ask questions about it. Any questions that I have asked have been answered to my satisfaction. I would like be a part of this study. I have been offered a copy of this Consent Form.

| Participant Signature | Date |
|-----------------------|------|
| If illiterate | |

| | e, this person should be selected by the participant and m). Participants who are illiterate should include their |
|---|---|
| · · | the consent form to the potential participant, and the estions. I confirm that the individual has given consent |
| Witness name and signature Da | te Thumb print of participant |
| maybe taken from you if you are hospital health. If there is anything left over after veryour permission to keep the leftover blood be useful for future research. Your specint testing for 10 years with your study ID information from the study; however, you research to be done on your blood and/or contract the study of the study in the study is the study of the study. | after CrAg testing and leftover cerebrospinal fluid that lized will be used to perform other tests about your we have done the required tests, we would like to ask and cerebrospinal fluid (CSF). These specimens could nens will be securely stored at the NHTD for future so that the specimen can be linked to your clinical ar name will not be on the specimens. The specific erebrospinal fluid will relate to HIV or other infections on private, your blood will be labeled with a code, and |
| future. No matter what you decide, it will | cerebrospinal fluid to be stored for possible use in the not affect whether you can be in the study, or your he statements below (or have them read to you) and |
| infections in people with HIV: \( \subseteq \text{Le} | g samples stored and used for future testing related to |
| Participant Signature | Date |

### **APPENDIX 4: ENROLLMENT FORM**

| Study ID | | of enrollment: | Data collector | |
|---|---|---|---|---|
| Ado | l sticker | or em omnene. | (Full name) | <del></del> |
| here | | / / | Signature | |
| | | · —— · ——— | <b>9</b> | <del></del> |
| I | I Socio - demographic information | | | |
| B01 | Sex | ☐1. Male ☐2. | . Female | |
| B02 | DOB | // | (dd/n | nm/yyyy) |
| | | 1. Single | | ☐4. Separated |
| B03 | Marital status | 2. Partnered | | 5. Divorced |
| | | ☐3. Married | | ☐6. Widowed |
| | | 1. No formal edu | ıcation | 5. Vocational |
| B04 | Education level (select the highest level attained) | 2. Primary school | ol(1st to 5th grade) | 6. University/College |
| | | 3. Secondary sch | nool(6 <sup>th</sup> to 9 <sup>th</sup> grade) | ☐7. Post graduate |
| | | 4. High school(10 <sup>th</sup> to 12 <sup>th</sup> grade) | | |
| | | 1. School/college | | 5. Agriculture/fishing |
| | | 2. Professional/o | | 6. Housewife |
| B05 | Occupation | 3. Shop worker/t | | 7. Retired |
| | | 4. Manual labour | | 8. Unemployed |
| | | 9. Other (specify | | |
| | | □1. ≤600,000VNI | | 4. >5,000,000-10,000,000VND |
| B06 | Monthly net income from all sources | <u></u> | 00,000VND | 5. >10,000,000 VND |
| | nom an sources | 3.>1,500,000-5 | ,000,000VND | |
| | Distance from home | ☐ 1. ≤5 km | 3. > 10 - 50 km | ☐ 5. >100 km |
| B07 | to clinic | □ 2. >5 – 10 km | $\Box$ 4. >50 – 100 km | 1 |
| | At the point of | 1. Yes (enrolled | during hospitalizatio | n) |
| B77 | enrolment, is the patient hospitalized? | ☐2. No (enrolled f | from OPC) | |
| | Does the patient have | □1. Yes | | |
| B78 | valid health insurance currently? | □2. No | | |

### **CRICS Study -** #4: Enrollment Form - Ver 2.1

| B79 | When did the patient register with the study clinic? | /(dd/mm/yyyy) |
|-----|------------------------------------------------------|---------------|
|-----|------------------------------------------------------|---------------|

| II | HIV Infection | | | | | |
|---|---|---|---|---|---|---|
| B08 | Blood specimen collection date for HIV confirmation testing(as written in the lab form presented by the patient) | | | /(dd/mm/yyyy) | | |
| B10 | The most recent CD | 04 count | | (cells/µL) | | |
| B11 | The most recent blo<br>specimen collection<br>count | | | //_ | (dd/mm/ <u>y</u> | уууу) |
| B81 | Check ALL OIs tha | t the patient has | in this vi | sit: | | |
| | Clinical stage 1 | Clinical stage 2 | 2 | Clinical sta | age 3 | Clinical stage 4 |
| | Asymptomatic Persistent generalized lymphadenopathy | body wt) Recurrent respiratory infe Papular prueruption | reight loss (<10% ody wt) Recurrent espiratory infections Papular pruritic | | loss >10% ht eary TB ained diarrhea endidiasis ained fever >1 especify | ☐ Extrapulmonary TB ☐ Pneumocystis pneumonia ☐ Oesaphogeal candidiasis ☐ CNS toxoplasmosis ☐ Other, specify ———— |
| Ш | Doct History | | | | | |
| 111 | Past History | | | | | |
| B16 | Diabetes | onfirmed | diagnosis | 2. Yes, self | f-report 3. No | |
| B17 | Hypertension | ☐ 1. Yes, c | onfirmed | firmed diagnosis 2. Yes, self-report 3. No | | |
| B18 | Kidney failure | ☐ 1. Yes, c | onfirmed | diagnosis | 2. Yes, self | f-report 3. No |
| B19 | Heart failure | ☐ 1. Yes, c | onfirmed | diagnosis | 2. Yes, self | f-report 3. No |
| B20 | Stroke | ☐ 1. Yes, c | onfirmed | diagnosis | 2. Yes, self | f-report 3. No |
| B21 | COPD | ☐ 1. Yes, c | onfirmed | diagnosis | 2. Yes, self | f-report 3. No |

| IV | <b>Current Symptoms</b> | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| B22 | Headache (Please circle the correct response) | C. | | ( ) | و ( المراق المرا | ,<br>((,)) | | (4.)<br>5 |
| B23 | Seizure | 1. Y | l'es | | ] 2. No | | 9. Not a | ssessed |
| B24 | Night sweat | <u> </u> | Yes | | ] 2. No | | 9. Not a | ssessed |
| B25 | Vomiting | <u> </u> | Yes | | ] 2. No | | 9. Not a | ssessed |
| B26 | Nausea | <u> </u> | Yes | | ] 2. No | | 9. Not a | ssessed |
| B27 | Abdominal pain | <u> </u> | Yes | | ] 2. No | | 9. Not a | ssessed |
| B28 | Constipation | <u> </u> | Yes | | ] 2. No | | 9. Not a | ssessed |
| B29 | Diarrhea | <u> </u> | Yes | | ] 2. No | | 9. Not a | ssessed |
| B30 | Cough | <u> </u> | Yes | | ] 2. No | | 9. Not a | ssessed |
| B31 | Dyspnea | <u> </u> | Yes | | ] 2. No | | 9. Not a | ssessed |
| B32 | Blurred vision | <u> </u> | Yes | | ] 2. No | | 9. Not a | ssessed |
| B33 | Skin rash | <u> </u> | Yes | | ] 2. No | | 9. Not a | ssessed |
| B34 | Fever | <u> </u> | Yes | | ] 2. No | | 9. Not a | ssessed |
| B35 | Photophobia | <u> </u> | Yes | | ] 2. No | | 9. Not a | ssessed |
| V | Physical Examination | ì | | | | | | |
| B36 | Glasgow score (3-15) | | | B37 | PR (bpn | n) | | |
| B38 | BP (mmHg) | | /_ | | | | | |
| B39 | Temperature (°C) | | | B40 | Weight | (kg) | | |
| B41 | RR (/min) | | | B42 | Height ( | (cm) | | |
| B43 | Chest examination(hea | | 1. Norrecify:_ | mal [ | ]2. Abnor | mal. | | |
| B44 | Abdominal examination | | | | | | | |
| B45 | Neurologic examination | examination 1. Normal 2. Abnormal, specify: 2.1. Neck stiffness 2.2. Kernig's sign 2.3. Cranial nerve paralysis 2.4. Hemiparesis 2.5. Other, specify: | | | | | _ | |
| B46 | Visual examination | | ☐ 1. Normal ☐ 2. Decreased ☐ 3. Fingers counting ☐ 4. Hand motion ☐ 5. Light perception ☐ 6. No light perception | | | | | |

### **CRICS Study -** #4: Enrollment Form – Ver 2.1

| ☐0. Fully active, able to carry on all pre-disease performance without restriction |
|---|
| 1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work |
| 2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours |
| ☐ 3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours |
| 4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair |

| VI | Lab Tests(Most recei | Date of testing (dd/mm/yy) | | | |
|---|---|---|---|---|---|
| 6.1 | Full Blood Count | Result | Unit | | // |
| B48 | Hemoglobin | | ☐(g/L)<br>☐(g/dL) | □Not available | |
| B49 | Leukocyte count | | (G/L) | ☐Not available | |
| B50 | Platelet count | | (G/L) | ☐Not available | |
| B51 | Neutrophil (%) | | % | ☐Not available | |
| B52 | Lymphocyte (%) | | % | ☐Not available | |
| 6.2 | Biochemistry | Result | | | / |
| B53 | Serum creatinine | | □μmol/L<br>□mg/dL | □Not available | |
| B54 | Serum urea | | □mmol/L □mg/dL | □Not available | |
| B55 | Serum glucose | | □mmol/L □mg/dL | □Not available | |
| B56 | AST/SGOT | | (U/L) | ☐Not available | |
| B57 | ALT/SGPT | | (U/L) | ☐Not available | |
| B58 | Total protein | | ☐ g/L<br>☐g/dL | □Not available | |
| B59 | Serum albumin | | □g/L<br>□g/dL | Not available | |

### **CRICS Study -** #4: Enrollment Form - Ver 2.1

| B60 | Serum bilirubin, total | | □μmol/L | Not available | |
|---|---|---|---|---|---|
| | | | mg/dL | | |
| 6.3 | Immunology | Result | | | |
| B61 | HBsAg | 1. Negativ | e <u>2. P</u> | ositive [ | 9. Not available |
| B62 | Anti-HCV | 1. Negativ | re <u></u> | ositive [ | _9. Not available |
| VII | Cryptococcus Antiger | n (CrAg) Test | Results | | |
| B14 | The date of OPC receive from the laboratory (do | | ılt | // | |
| B15 | CrAg result? | | □ 1. Ne | egative <b>\rightarrow End</b> | 2. Positive |
| | , | | | | |
| B63 | Patient is female and Patient is male or fer Date of last normal mer period | • | | | |
| B64 | Pregnancy test | | 1. Negative | 2. Positive | 9. Not done |
| B65 | Was fluconazole started (current visit)? | , , , | 1. Yes<br>→Go to B75 | | specify the reason |
| B75 | Date of starting flucona | - | /<br>→ Complete F | /(dd | /mm/yyyy)<br><b>(ppendix 19)</b> |
| B73 | Hospitalization for lum | | <u> </u> | | |
| B74 | Name of the hospital | | | | |

**Date of enrollment:** 

**Study ID** 

Other drugs

1.2

#### **APPENDIX 5: STARTING ART FORM**

(These data should be transcribed from clinical notes and pharmacy prescriptions whenever ART is initiated)

**Data collector** 

| Add sticker<br>here | | | (Full name) Signature |
|---|---|---|---|
| I | Treatment | t Information | |
| 1.1 | Opportun | istic Infection Prevention and Tr | eatment |
| X01 | Is the patie | ent on cotrimoxazole prophylaxis? | <ul><li>☐1. Yes</li><li>☐2. No → Skip to X14</li></ul> |
| X01a | Date of sta | rting cotrimoxazole prophylaxis | // |
| X01b | Cotrimoxa | zole dose per day? | ☐1. 480 mg/ tablet x tablet ☐2. 960 mg/ tablet x tablet |
| X14 | Is the patie | ent on anti-TB medication? | □1. Yes □2. No <i>→Skip to X15</i> |
| X14a | Current TE record)s | 3 regimen (verify from the patient | ☐ SRHZE ☐RHZE ☐RHE ☐RH ☐ ZEK <sub>m</sub> (C <sub>m</sub> )L <sub>fx</sub> P <sub>to</sub> C <sub>s</sub> (PAS) ☐ ZEL <sub>fx</sub> P <sub>to</sub> C <sub>s</sub> (PAS) ☐ Other: ☐Unknown |
| X14b | Starting da | te of current TB regimen | //Unknown |
| X14c | Number of | anti-TB tablets taken each day | tablets_Unknown |
| X15 | Is the patient on Isoniazid prophylaxis? | | <ul><li>☐1. Yes</li><li>☐2. No →Skip to X02</li></ul> |
| X15a | If yes, start | ting date? | //Unknown |
| X15b | Number of | isoniazid tablets per day | tablets |

### CRICS Study - #5: Starting ART Form Ver 2.1

| X02 | Is the patient on other medications(besides anti-TB drugs, Cotrimoxazole, Isoniazid and ARVs) | | <ul> <li> □ 1. Yes □ 2. No → Skip to 1.3 </li> </ul> | | | |
|---|---|---|---|---|---|---|
| | | OTHER<br>DRUG1 | OTHERD<br>RUG2 | OTHERD<br>RUG3 | OTHER<br>DRUG 4 | OTHERD<br>RUG 5 |
| X04 | Name of drug | | | | | |
| X04a | Number of tablets per day | | | | | |
| 1.3 | ART treatment at current visit | t | | | | |
| X08 | Date ART started | / | / | (dd | /mm/yyyy) | |
| X16 | Dose adjustment for kidney failure patients | ☐ 1. Yes ☐ 2. No | | | | |
| | ARV regimens (Dosage) | TDF + | | | | |
| X17 | | AZT + | 3TC | + E | FV | |
| | | AZT + | | | VP | |
| X18 | Total number of all ARV | + | | + _ | | |
| Alo | tablets taken per day | | table | ets | | |

### CRICS Study- #6 Follow-up form - Ver 2.1

| Time of visit: _ |
|------------------|
|------------------|

### **APPENDIX 6: FOLLOW-UP FORM**

| Subje | ect ID | Date of Visit: | Data Collector<br>(Name) – | |
|---|---|---|---|---|
| | Add sticker<br>here | / | Signature _ | |
| | Visit type (according to appointments) | | ointment <del>&gt;</del> Complete Appendix<br>e, Missed Appointment Form in<br>rm | |
| I | HIV Infection | | | |
| D0A | Does the patient h | ave health insurance? | ☐ 1. Yes☐ 2. No | |
| B77 | At the point of enhospitalized? | rollment, is the patient | ☐1. Yes (enrolled during ☐2. No (enrolled from OF | - , |
| B79 | When did the pati study clinic? | ent register with the | /(d | d/mm/yyyy) |
| D01 | Latest test CD4 result (cells/µL) | | (cells/μL) No result since the last | testing → Skip to D03 |
| D02 | Date of latest CD4 testing (check CD4 result form for date) | | // | (dd/mm/yyyy) |
| D63 | Check ALL OIs the | nat the patient has in this | visit: | |
| | Clinical stage 1 | Clinical stage 2 | Clinical stage 3 | Clinical stage 4 |
| | Asymptomatic Persistent generalized lymphadenopathy | weight loss (<10% body wt) | <ul> <li>Weight loss &gt;10%</li> <li>body weight</li> <li>Pulmonary TB</li> <li>Unexplained diarrhea</li> <li>&gt;1 month</li> <li>Oral candidiasis</li> <li>Unexplained fever &gt;1 month</li> <li>Other, specify</li> </ul> | ☐ Extrapulmonary TB ☐ Pneumocystis pneumonia ☐ Oesaphogeal candidiasis ☐ CNS toxoplasmosis ☐ Other, specify ———— |
| D05 | Latest viral load r | esult (copies/ml) | (copies/ml) [ ] 1 | Not done <b>→Skip to D23</b> |
| D06 | Latest date of test<br>(dd/mm/yy) | ing viral load | / | |
| II | Hospitalization | | | |
| D23 | Was the patient l | nospitalized 🗀 Ves | 2 | |

### CRICS Study-#6 Follow-up form - Ver 2.1

| | since the last visit for CRICS data were coll | | <u></u> | 2. No <b>→Go to D40</b> | | | | |
|---|---|---|---|---|---|---|---|---|
| D23A | Total number of hospitalizations since visit for which CRICS were collected? | | | (times) ->Complete Hospitalization Form for a not completed | | | any hospi | talizations if |
| III | Physical Examination | on | | | , | | | |
| D40 | Glasgow score (3-15)(see Appendix) | _ | D41 | Temperature (°C) | | D42 | Weight | (kg) |
| D43 | Neurologic examination | <u>1</u> . | No me | eningeal signs 🔲 | 2. Meninge | al signs | s found | |
| D62 | 1. Restricted in pholight or sedentary nate 2. Ambulatory and and about more than 3. Capable of only hours | <ul> <li>□ 0. Fully active, able to carry on all pre-disease performance without restriction</li> <li>□ 1. Restricted in physically strenuous activity but ambulatory and able to carry out work of light or sedentary nature, e.g., light house work, office work</li> <li>□ 2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours</li> <li>□ 3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours</li> <li>□ 4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair</li> </ul> | | | | ivities. Up<br>waking | | |
| IV | Lab Tests (The most i | recent if r | ot rec | orded in the last | CRICS vi | isit)) | Date | e of testing |
| · | <ul><li>☐1. Yes</li><li>☐2. No → Skip to D5.</li></ul> | | | | | , , | | 8 |
| 5.1 | Full Blood Count | Res | sult | Unit | | | /_ | / |
| D44 | Hemoglobin | | | ☐(g/L)<br>☐(g/dL) | □Not ava | ailable | | |
| D46 | Platelet count | | | (G/L) | ☐Not ava | ailable | | |
| 5.2 | Biochemistry | Result | | Unit | | | /_ | / |
| D49 | Serum creatinine | | | □μmol/L<br>□mg/dL | □Not ava | ailable | | |
| D51 | AST/SGOT | | | (U/L) | ☐Not ava | ailable | | |
| D52 | ALT/SGPT | | | (U/L) | ☐Not ava | ailable | | |

### CRICS Study- #6 Follow-up form - Ver 2.1

| VI | Anti-retroviral Thera | py (ART) | | | |
|---|---|---|---|---|---|
| D53 | Is patient on ART? | 2. Has not be 3. Starting A | <ul> <li>☐ 1. Being treated</li> <li>☐ 2. Has not been treated yet →Skip to VII. Current symptoms</li> <li>☐ 3. Starting ART at this visit →Skip to VII. Current symptoms and complete Form 05: Starting ART form</li> </ul> | | |
| D24 | Common ARV side effects | ☐1. Yes. If y ☐2. No | es, sp | pecify | → Complete Form 09: AE |
| D61 | Current ART regimen | 1. Continue 2. Switched another regime (specify below | to<br>en | 1. TDF + 3 2. TDF + 3 3. TDF + 3 4. AZT + 3 5. AZT + 3 | TC + EFV TC + NVP TC + LVP/r TC + EFV TC + EFV TC + NVP |
| D61a | Date of switching ART | regimen | | / | /(dd/mm/yy) |
| D61b | Reason for changing regimen | 1. Intolerance 2. Treatment 3. Other, specific | t failı | | |
| 6.1 | ART Adherence | | | | |
| D54 | Adherence based on times medications missed | ☐ 1. Good (≤ ☐ 2. Average ☐ 3. Bad (> 8 | (4-8 1 | times/month) | 4. Not assessed If no assessment, please specify the reason: |
| D55 | Thinking about the pass average, how would yo ability to take all your prescribed? | ou rate your | | . Very poor<br>. Poor<br>. Fair | |
| D57 | Since the last visit, hav missed a dose of antire medicines? | | | . Yes<br>. No <b>→ Skip to</b> | D D 58 |
| D58 | Visual analogue scale f<br>adherence (Show the pa<br>scale and ask the patien<br>adherence) | atients the VAS | Sco<br>If th | | Ag-negative <b>→ End</b> |

| FOR CRAG-POSITIVE ONLY | | | | | | | |
|---|---|---|---|---|---|---|---|
| D64 | Current place of residence | | | | | | |
| VII | Current Sympto | ms (the timing of the | e closest exa | mination)fo | or CrAg + | only | |
| | Symptoms | Present | (ON | LY RECORD<br>EATED WIT<br>SYMF<br>2.<br>Unlikely<br>related | D IF THE P | PATIENT IS<br>NAZOLE an | BEING |
| D08 | Headache | ☐ 1. Yes ☐ 2. No | | | | | |
| D09 | Seizure | ☐ 1. Yes ☐ 2. No | | | | | |
| D10 | Night sweat | ☐ 1. Yes ☐ 2. No | | | | | |
| D11 | Vomiting | ☐ 1. Yes ☐ 2. No | | | | | |
| D12 | Nausea | ☐ 1. Yes ☐ 2. No | | | | | |
| D13 | Abdominal pain | ☐ 1. Yes ☐ 2. No | | | | | |
| D14 | Constipation | ☐ 1. Yes ☐ 2. No | | | | | |
| D15 | Diarrhea | ☐ 1. Yes ☐ 2. No | | | | | |
| D16 | Cough | ☐ 1. Yes ☐ 2. No | | | | | |
| D17 | Dyspnea | ☐ 1. Yes ☐ 2. No | | | | | |
| D18 | Blurred vision | ☐ 1. Yes ☐ 2. No | | | | | |
| D19 | Skin rash | ☐ 1. Yes ☐ 2. No | | | | | |
| D20 | Fever | ☐ 1. Yes ☐ 2. No | | | | | |
| D21 | Photophobia | ☐ 1. Yes ☐ 2. No | | | | | |
| VIII | Pregnancy test a | nd Fluconazole Ther | apy for Cra | Ag (+) patie | ents only | | |
| | ☐ Patient is male or female but menopausal or over 55 years old → Skip to D30 ☐ Patient is female and of reproductive age → Go to D25 | | | | | | |
| D25 | Pregnancy □Pregnancy was not diagnosed in the last visit →Go to D25a □Pregnancy was diagnosed in the last visit, note pregnancy status since then →Go to D25b | | | | | | |
| D25a | 1.Date of last normal menstrual period//(dd/mm/yy) If the patient does not remember, estimate last normal menstrual period// (dd/mm/yy) Over 5 weeks →Do pregnancy test and record results of the test below | | | | | | |

☐Under 5 weeks → Skip to D30  $\Box$ Do not know → *Skip to D30* 

### CRICS Study- #6 Follow-up form - Ver 2.1

| | 3. Pregnancy test | 1. Positive 2. Negative | e 3. Not done |
|---|---|---|---|
| D25b | 1. Healthy pregnancy | | |
| | 2. Spontaneous abortion | Specify date (dd/mm/yy): | // |
| | 3. Medical abortion | Specify date (dd/mm/yy): | // |
| | | 4a. Specify date | //(dd/mm/yy) |
| | 4. Gave birth | 4b. Congenital abnormality | □1. Yes □2. No |
| | Fluconazole Adherence | | |
| D30 | During the past 4 weeks, | ☐1. Very poor | ☐5. Very good |
| | basically how would you rate | □2. Poor | ☐6. No assessment, please |
| | your ability to take all your | ☐3. Fair | specify the reason: |
| | medications as prescribed? | ☐4. Good | |
| D32 | Since the last attended scheduled | visit, have you ever missed a | □1. Yes |
| | dose of fluconazole? | | 2. No <b>→ Go to D33</b> |
| D31 | During the past 4 days, how many | times have you missed taking | (times) |
| | your medication (fluconazole)? (n | umeric response) | () |
| D33 | Visual analogue scale for fluconaz | zole adherence (Show the | Score: |
| | patients the VAS scale and ask the | patient to rate their | |
| | adherence) | | |
| | <del>-</del> | | |

#### **APPENDIX 7: HOSPITALIZATION FORM Study ID** Data collector **Date of collection:** (full name) Add sticker Signature here \_\_\_\_/ \_\_\_\_/ I **Information about Hospitalization** Source of information E0 Hospital chart (Check all that apply) Discharge certificate provided to patient Discharge summary provided to OPCs Communication with hospital clinicians Patient self-reported No information -> End of the form E01 Date of admission (dd/mm/yyyy) E02 Date of discharge (dd/mm/yyyy) E03 Name of the hospital E05 Discharge diagnosis 1. Cryptococcal meningitis 2. ART adverse reaction 3. Fluconazole adverse reaction 4. Opportunistic infections, specify: 9. Others, specify: E06 Patient's outcome at the time of 1. Fully recovered discharge 2. Partially recovered 3. Not recovered ☐ 4. Worsened $\Box$ 5. Dead → Complete Off-Study Form II **Clinical Signs and Laboratory Results Date of testing** E25 CD4 test done during current ☐1. Yes hospitalization $\square$ 2. No $\rightarrow$ Skip to E08 Unknown

### **CRICS Study -** #7 Hospitalization Form – Ver 2.1

| E07 | CD4 count results (from sample taken during current hospitalization) | | (c<br>]Not availab | ells/μL)<br>ble | / |
|---|---|---|---|---|---|
| E08 | Meningeal signs | | □1. Yes □ 2. No | | |
| | | | Unknown | | |
| E09 | Performing lumbar puncture? | | 1. Yes | | |
| | | | $\]$ 2. No $\rightarrow G$ | o to Part IV | |
| III | CSF Analysis Results | | | | |
| 3.1 | Cytology | | Date of tes | sting:// | (dd/mm/yy) |
| E10 | WBC | | | (cells/nm³) | □Not available |
| E11 | Neutrophils | | | % | ☐Not available |
| E12 | Lymphocytes | | | % | ☐Not available |
| 3.2 | Biochemistry | | Date of tes | sting:// | (dd/mm/yy) |
| E13 | CSF glucose | | | □ μmol/L<br>□ mg/dL | ☐Not available |
| E14 | CSF protein | | | ☐ g/L | ☐ Not available |
| | | | | □g/dL | Not available |
| E15 | Pandy reaction | | □1. Positi | ve 2. Negative | 9. Not available |
| 3.3 | Microbiology | | | | |
| E16 | Indian ink stain | | □1. Positi | ve 2. Negative | 9. Not available |
| E17 | CSF CrAg | | 1. Posit | ive 2. Negative | ☐9. Not available |
| E26 | CSF culture for bacteria | | □1. Positi | ve, specify: | |
| | | | ☐2. Negat | rive | |
| | | | 9. Not a | vailable | |
| E27 | CSF culture for fungi | 1. Positive, specify: | | | |
| | | 2. Negative | | | |
| | | | 9. Not a | | |
| IV | Antifungal therapy for cryptoco | occa | l meningitis | | |
| D20 | Is the patient being treated with antifungal drugs for | <u> </u> | Yes | | |
| | cryptococcal meningitis? | 2 | . No <b>→</b> <i>End</i> | | |

### **CRICS Study -** #7 Hospitalization Form – Ver 2.1

| E21 | Induction therapy | □1. Yes □2. No → | End | | |
|---|---|---|---|---|---|
| E22 | Regimen for induction therapy | Drugs | Dose<br>(mg/<br>day) | Date of starting (d/m/y) | Date of ending (d/m/y) |
| | | ☐1. Amphotericin B IV | | _/_/_ | _/_/_ |
| | | ☐2. Fluconazole IV | | // | // |
| | | ☐3. Flucytosine IV | | // | // |
| | | 4. Fluconazole PO | | // | _/_/_ |
| E23 | Consolidation therapy ☐1. Yes ☐2. No <b>→End</b> | Fluconazole PO | | _/_/_ | // |
| E24 | Maintenance therapy ☐1. Yes ☐2. No → End | Fluconazole PO | | _/_/_ | // |

### **APPENDIX 8: LATE ATTENDANCE, MISSED APPOINTMENT FORM**

| Subject ID | | <b>Data Collector</b> |
|-------------|----------------|-----------------------|
| Add sticker | Date of visit: | (Name) |
| here | / / | Signature |

| | Late Attendance, Missed Appointment | |
|---|---|---|
| L1 | Today's date (dd/mm/yy) | // |
| L2 | Date of patient's original appointment(dd/mm/yy) | /// |
| L4 | Number of phone calls before patient was successfully contacted | |
| | | times |
| L5 | Number of home visits done before patient was successfully contacted | times |
| L6 | What was the main reason for missing original appointment | <ul> <li>☐ 1. Forgot</li> <li>☐ 2. Not had enough pills</li> <li>☐ 3. Did not have money for transport</li> <li>☐ 4. Had family emergency</li> <li>☐ 5. Was away traveling</li> <li>☐ 6. Could not get time off work</li> <li>☐ 7. Other, specify</li> </ul> |

#### **APPENDIX 9: AE REPORTING FORM**

**Vietnam Cryptococcal Retention in Care Study (CRICS)** 

| Add | sticker |
|------|---------|
| here | |

| Date of reporting:/ | |
|---|---|
| Name of reporter: | |
| Did the patient have any unexpected adverse event (AE) in this study? | ☐ No (If yes, please list all adverse events in the below table) |

| Level 1 = Slightly 2 = Moderatel y 3 = Severely | Related to fluconazole? 0 = Not related: clearly explained by another, documented cause 1 = Unlikely related: more likely explained by a cause other than fluconazole 2 = Possibly related: may be related to the drug or to another cause 3 = Probably related: more likely related to the drug than to another cause 4 = Definitely related: direct association with fluconazole | Applied management related to fluconazole 1 = Not available 2 = Stop using fluconazole permanently 3 = Stop using fluconazole temporarily 4 = Reduce dose 5 = Increase dose 6 = Delay | Adverse event's outcome (AE) 1 = Stabilization, no complication 2 = AE is still happening - no therapy 3 = AE is still happening- being treated 4 = Still happening - not treated 5 = Still happening - was treated 6 = Death 7 = Do not know (lost to follow-up) |
|---|---|---|---|
|---|---|---|---|

# Serious adverse event? (If yes, complete serious adverse event form -SAE)

- Death
- Life-threatening event
- Hospitalization, prolongation of existing hospitalization, or rehospitalization.
- Persistent or significant disability/incapacity
- An important medical event.
- Pregnancy in a woman taking fluconazole
- A congenital abnormality or spontaneous abortion

### CRICS Study-#9 AE Reporting Form - Ver2.1

| Adverse events relatedness to fluconazole | Date of starting | Level | Relatedness<br>to<br>fluconazole | Management | Adverse event's outcome | Serious adverse event? |
|---|---|---|---|---|---|---|
| 1. | | | | | | ☐Yes ☐ No |
| 2. | | | | | | ☐Yes ☐ No |
| 3. | | | | | | ☐Yes ☐ No |
| Other unexpected adverse events | | | | | | |
| 1. | | | | | | |
| 2. | | | | | | |
| 3. | | | | | | |
| Narrative Summary of AE: | | | | | | |

CRICS Study- #10A: SAE Reporting Form - Ver 2.1

#### **APPENDIX 10A: SAE REPORTING FORM (SAE)**

(Based on Serious adverse events form attached to Official Dispatch No. 6586/BYT-K2DT dated 02/10/2012)

| ☐ Initial Report ☐ Follow - up report (time ☐ Final report |
|------------------------------------------------------------|
| f death |
| nce |
| n's |
| in 🔲 |
| _ |

| CRICS Study-#10A: SAE Reporting Form - Ver 2.1 |
|---|
| <b>7</b> |
| Pre-clinical tests: |
| Why the researcher identified this is SAE: |
| Relatedness of SAE to fluconazole (as identified by researcher) |
| Unrelated: clearly explained by another, documented cause |
| Unlikely related: more likely explained by a cause other than fluconazole |
| Possibly related: may be related to the drug or to another cause |
| ☐ Probably related: more likely related to the drug than to another cause |
| Definitely related: direct association with fluconazole |
| This SAE is: Expected |
| ☐ Unexpected |
| (The nature, frequency and severity of adverse events in the document on product research/literature |
| or have observed or not) |
| □Yes→ Expected □No→ Unexpected |
| Severity of SAE: |
| Death |
| Life – threatening |
| ☐ Not cause death or life – threatening (specify) |
| 3. Information about treatment/management SAE |
| The simultaneous drugs before appearing SAE |
| Drugs, medical interventions have been done to manage the study subject with SAE (specify) |
| TI '4 4' C 4 1 1' 4 '4 CAE' 4 4 4 4' 1' 1 |
| The situation of study subject with SAE in the current reporting period |
| Not recovered Recovered with sequelae Death |
| Being recovered Recovered without sequelae Unclear |

| CRICS Study-#10A: SAE | Reporting Form - Ver 2.1 | | |
|---|---|---|---|
| 4. Professional comments | of local IRB/scientific coun | cil/research chair | unit |
| Suggestions: | | | |
| For study subject: | Continuing study | ☐ Stopping | ☐ Withdrawing from |
| | | temporary | the study |
| For study: | Continuing study | ☐ Stopping temporary | ☐ Withdrawing from the study |
| 5. Principal investigator's | suggestions | | |
| Reporter (signature and mark | k, occupational skills) | | |
| Head of Unit (signature and r | nark) | | |

#### **APPENDIX 10B: CLINICAL STUDY SAE REPORT FORM**

| Report classification | ☐ Initial report | | | | | |
|---|---|---|---|---|---|---|
| | Follow up report | <b>#</b> 1 | <b>#</b> 2 | <u></u> #3 | <b>#4</b> | Last report |
| Date of report:/(dd/m | | | | | | |
| 1. Subject information | | | | | | |
| Study ID | | Study | site (region | ): | | |
| Gender | | D.O.B | | | | / |
| Date of enrollment | / | CD4 r | esult at enro | ollment | · | |
| Serum CrAg testing | ☐ Positive ☐ Negative | Date of | f HIV conf | irmation | /_ | / |
| WHO clinical stage at enro | olment: | WHO | clinical stag | ge at the ti | ime of th | e report: |
| OIs that imply above WHO | O clinical stage: | OIs th | at imply abo | ove WHO | clinical | stage: |
| 2. SAE information | | • | | | | |
| Serious adverse event | | | | | | |
| Date of occurrence | / | | Date of n | otification | 1 | |
| Alternative causality | | | Specify: | | | |
| 3. Event description | | | | | | |
| | Descriptions | Source of information | | | If other, specify or comment | |
| Sign and symptoms | | | | | | |
| Progression | | | | | | |
| Possible causes/diagnosis | | | | | | |
| Treatment/management | | | | | | |
| 4. Additional information: | | | | | | |

### 5. Additional information for CrAg (+) patients:

| Treatment | | Date start | Date end |
|---|---|---|---|
| Amphotericin B | Yes | / | / |
| | ☐ No | | |
| Study Fluconazole – induction phase (900 | Yes | / | / |
| mg/day) | ☐ No | | |
| Study Fluconazole – consolidation phase | Yes | / | / |
| (450 mg/day) | ☐ No | | |
| Study Fluconazole – maintenance phase | Yes | / | [6 months after CD4 >200] |
| (150-200 mg/day) | ☐ No | | |
| Fluconazole (150mg)- maintenance phase | Yes | / | / |
| upon the complement of 12 month study | ☐ No | | |
| follow-up (based on treating doctor's judgement) | | | |

#### 6. Additional information for case of deaths:

| If the patient died, specify the place of death: Home Hospital Other | | If other, specify: | |
|---|---|---|---|
| If the patient died at home, was the patient discharged | from hospital for palliative | care within 7 days before death: Y | es No. If yes: |
| Date of hospitalization:// | | Hospital name: | |
| Date of discharge:/ | | Diagnosis on admission: | |
| Cause of death: | Specify/comments | How were causes of death determined | Confirmatory diagnostics were performed |
| Primary cause: | | | □No |
| | | | Yes. If yes, specify: |
| Underlying cause 1: | | | □No |
| | | | ☐ Yes. If yes, specify: |
| Underlying cause 2: | | | □No |
| | | | ☐ Yes. If yes, specify: |
| Specify OIs (using WHO AIDS-defining illness list) | | | □No |
| at the time of death: | | | ☐ Yes. If yes, specify: |
| Was death related to Cryptococcus infection? | □ No | If yes, specify how determined: | □ No |
| | Yes. | 70.1 | Yes. |
| | | If other, specify: | If yes, specify: |
| | 1 1 1111 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | |
| Underlying diseases or comorbidity at the time of deat | h in additional to HIV: | | |

#### CRICS Study-#10B: Clinical Study SAE Report Form - Ver 2.1

#### Does SAE related to study fluconazole?

| Yes | ☐ No | Not related: clearly explained by another, documented cause |
|---|---|---|
| Yes | ☐ No | Unlikely related: more likely explained by a cause other than fluconazole |
| Yes | ☐ No | Possibly related: may be related to the drug or to another cause |
| Yes | ☐ No | Probably related: more likely related to the drug than to another cause |
| Yes | ☐ No | Definitely related: direct association with fluconazole |
| 7. Action | - | |

| ☐ Follow-up |
|-------------|
|-------------|

☐ No action required

#### 8. Relevant investigation data

(Recorded if the test results are within two weeks since the date of death)

| Test | Unit | Date | Result | Note |
|----------------------|--------|------|--------|-----------------|
| Complete Blood Count | | // | | ☐ Not available |
| WBC | K/µL | | | _ |
| Neutrophils | % | | | _ |
| Lymphocytes | % | | | _ |
| RBC | M/μL | | | _ |
| НСВ | g/dL | | | _ |
| PLT | K/µL | | | _ |
| Biochemistry | | / | | ☐ Not available |
| Creatinine | μmol/L | | | _ |
| Urea | mmol/L | | | _ |
| Glucose | mmol/L | | | _ |
| AST/SGOT | U/L | | | _ |
| ALT/SGPT | U/L | | | _ |
| Total protein | g/L | | | _ |
| Albumin | g/L | | | _ |
| Total Bilirubin | μmol/L | | | _ |
| CSF analysis | | // | | ☐ Not available |
| Cell count | | | | _ |
| Cell differential | | | | _ |
| Protein | g/L | | | _ |
| Glucose | mmol/L | | | _ |
| Radiology | | | | ☐ Not available |

CRICS Study-#10B: Clinical Study SAE Report Form - Ver 2.1

| Test | | Unit | Date | Result | Note |
|--------------|-----------------|------|------|--------|-----------------|
| Ultrasound | Abdomen | | | | ☐ Not available |
| | GeneXpert | | // | | ☐ Not available |
| Microbiology | Hepatitis virus | | | | ☐ Not available |
| | Fungal test | | // | | ☐ Not available |
| Other: | | | // | | ☐ Not available |

### **APPENDIX 11: OFF-STUDY FORM**

| Subject ID Add sticker here | | Date of Collec | tion | On (Name) ———————————————————————————————————— |
|---|---|---|---|---|
| | | / | | Signature |
| F01 | | going Off-Study | 2. Lost to for 3. Withdrey | ed study $\Rightarrow$ Skip to F08 collow-up $\Rightarrow$ Skip to F05 ew consent $\Rightarrow$ Skip to F08 red out $\Rightarrow$ Skip to F08 electify: |
| If the reason for off-study is Death (5) | | | | |
| F02<br>F03 | Date of death (dd/mm/yyyy)// Cause of death 1. Confirmed cryptococcal meningitis 2. Suspected cryptococcal meningitis 3. Opportunistic infection, specify: 4. Unknown 5. Addiction due to overdose 9. Others, specify | | | F03A. Source of death causes report Hospital's death documents/medical record Communication with treating doctor Reported by patient's family |
| F04 | Location of | □ 1. Home □ 2. Hospital □ 9. Others, s | | pecify: |
| F05 | death (withi | as patient hospitalized before ath (within 1 week before the ath occurred) 1. Yes → Complete Hospitalized before 2. No → End | | nplete Hospitalization Form if not recorded |
| If the reason for off-study is Lost to follow-up (2) | | | | |
| F05 | Date of last with patient | attempt to contact | / | /(dd/mm/yyyy) |
| F06 | Method last patient | used to try to contact | 1. Three att | |

### CRICS Study-#11: Off-study Form - Ver 2.1

| F07 | Patient's statu | | 1. Alive 2. Dead 9. Unknown Idy (1), Withdraw consent (3), or Transferred out (4) |
|---|---|---|---|
| F08 | Outcome<br>scale<br>(explanation<br>of activity) | □ 0. Fully active, able to carry on all pre-disease performance without restriction □ 1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work □ 2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours □ 3. Capable of only limited self-care, confined to bed or chair more than 50% of waking hours □ 4. Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair | |
| If the patient returns to the initial OPC and continue take part in the study after having been lost to follow-up, Withdraw consent, or Transferred out | | | |
| F09 | Date of return | Patient's new OPC ID: Patient's previous OPC | |
# APPENDIX 12: CLINICAL SCORING TOOLS AND WHO CLINICAL STATING OF HIV/AIDS

### Sub-Appendix 1: Visual Analogue Scale (VAS) for Pain Assessment

To assess the severity of pain, a six-level VAS tool is utilized. This VAS has been included in the CRFs. Following is the definition of each level of pain severity.



# Score Definition of pain severity 0 No pain at all 1 Very mild pain 2 Mild pain 3 Moderate pain 4 Very severe pain 5 The worst pain ever

### Sub-Appendix 2: Visual Analogue Scale (VAS) for Adherence

To assess ART and fluconazole adherence, a VAS tool is utilized in combination with other measures. The following VAS is to show the data collector how to use this tool. A large version printed in a plastic-wrapped A4-sized paper is used during interviewing the patient for their adherence.



Ask the patient: to think back over the past month and identify the times when he or she either missed a dose or took it at the wrong time. Show the patient this VAS. Tell the patient that if he/she had taken all medicine doses, he/she would point to 10 (biggest round); and if he/she had missed all the doses, he/she would point to 0 (no round). Now give the patient an opportunity to point out their level of adherence. Write the score in the blank.

### CRICS study - #12 Clinical scoring tools and WHO clinical stating of HIV/AIDS - Ver 2.1

### **Sub-Appendix 3: Glasgow coma scale**

| Category | Response | Grade |
|----------|-------------------------------------------|-----------|
| Eyes | Opens eyes spontaneously | 4 |
| | Opens eyes in response to speech | 3 |
| | Opens eyes in response to painful stimuli | 2 |
| | Does not open eyes | 1 |
| Motor | Obeys | 6 |
| | Localize | 5 |
| | Withdrawal | 4 |
| | Abnormal flexion | 3 |
| | Abnormal extension | 2 |
| | No motor response | 1 |
| Verbal | Orientated | 5 |
| | Confused (Disoriented) | 4 |
| | Inappropriate words | 3 |
| | Incomprehensive sounds | 2 |
| | No response 1 | 1 |
| | Total: | 15 points |

### Assess the severity of a brain injury using Glasgow coma scale:

15 points: Normal

9-14 points: Light unconsciousness6-8 points: Heavy unconsciousness

4-5 points: Deep coma

1-3 points: Very deep coma, very poor chance of recovery

### Sub-Appendix 4: WHO clinical staging of HIV disease in adults and adolescents

# Clinical stage 1 Asymptomatic or Persistent generalized lymphadenopathy Clinical stage 2 Moderate unexplained weight loss (<10% of presumed or measured body weight) Recurrent respiratory tract infections (sinusitis, tonsillitis, otitis media, pharyngitis) Herpes zoster Angular cheilitis Recurrent oral ulceration Papular pruritic eruption Fungal nail infections Seborrheic dermatitis Clinical stage 3

### CRICS study - #12 Clinical scoring tools and WHO clinical stating of HIV/AIDS - Ver 2.1

Unexplained severe weight loss (>10% of presumed or measured body weight)

Unexplained chronic diarrhoea for longer than 1 month

Unexplained persistent fever (intermittent or constant for longer than 1 month)

Persistent oral candidiasis

Oral hairy leukoplakia

Pulmonary tuberculosis

Severe bacterial infections (such as pneumonia, empyema, pyomyositis, bone or joint infection, meningitis, bacteraemia)

Acute necrotizing ulcerative stomatitis, gingivitis or periodontitis

Unexplained anaemia (<8 g/dl), neutropenia ( $<0.5 \times 10^9$ /l) and/or chronic thrombocytopenia ( $<50 \times 10^9$ /l)

### Clinical stage 4

HIV wasting syndrome

Pneumocystis (jirovecii) pneumonia

Recurrent severe bacterial pneumonia

Chronic herpes simplex infection (orolabial, genital or anorectal of more than 1 month's duration or visceral at any site)

Oesophageal candidiasis (or candidiasis of trachea, bronchi or lungs)

Extrapulmonary tuberculosis

Kaposi sarcoma

Cytomegalovirus infection (retinitis or infection of other organs)

Central nervous system toxoplasmosis

HIV encephalopathy

Extrapulmonary cryptococcosis, including meningitis

Disseminated nontuberculous mycobacterial infection

Progressive multifocal leukoencephalopathy

Chronic cryptosporidiosis

Chronic isosporiasis

Disseminated mycosis (extrapulmonary histoplasmosis, coccidioidomycosis)

Lymphoma (cerebral or B-cell non-Hodgkin)

Symptomatic HIV-associated nephropathy or cardiomyopathy

Recurrent septicaemia (including non-typhoid Salmonella)

Invasive cervical carcinoma

Atypical disseminated leishmaniasis

**CRICS study** - #13 Invitation to participate in Cryptococcal Antigen Screening Program - Ver 2.1

## APPENDIX 13: Invitation to participate in Cryptococcal Antigen Screening Program NHTD/TDH/CDC/VAAC

### **CRAG Screening Program**

RE: Invitation to participate in Cryptococcal Antigen (CrAg) Screening Program

Dear Dr.

In 2011, the World Health Organization (WHO) recommended that patients with low CD4 be screened for CrAg and, if positive, be preemptively treated with oral fluconazole before starting ART to reduce mortality from undiagnosed infection. In the same guidance, WHO recommends discontinuation of primary prophylaxis with fluconazole as an intervention in the prevention of cryptococcal meningitis (CM).CrAg screening has been shown to be cost-effective where the prevalence of CrAg positivity in persons living with human immunodeficiency virus (PLHIV) with CD4<100 cells/μL exceeds 0.6 to 3%, depending on the setting. The prevalence of CrAg in PLHIV in Vietnam is not clearly known. However a study conducted on archived specimens showed that the prevalence is 2% in the North and 6% in the South. The prevalence in the middle of Vietnam is not known. Information from this study will help the Vietnam Administration of HIV/AIDS Control (VAAC) decide whether to implement the WHO guidelines in Vietnam.

To this end, the National Hospital for Tropical Diseases (NHTD) in collaboration with the Tropical Diseases Hospital (TDH), the United States Centers for Disease Control and Prevention (CDC) and the VAAC is about to begin rollout of a program to screen PLHIV with CD4<100 for cryptococcal antigen. We want to know if the screening PLHIV with CD4<100 for cryptococcal disease using a lateral flow assay (LFA) and preemptively treating those who are CrAg-positive with oral fluconazole 900 mg daily for 2 weeks followed by a consolidation dose of 450 mg daily for 8 weeks, followed by 200 mg for maintenance reduces mortality and improves retention in care. We will also assess the costs associated with such screening at in Vietnam

To help VAAC and the Ministry of Health (MoH) rollout the intervention, we will ask clinics to start screening all patients with CD4  $\leq$  100 cells/ $\mu$ L for CrAg. Your clinic is one of those identified to participate in this evaluation.

**CRICS study** - #13 Invitation to participate in Cryptococcal Antigen Screening Program - Ver 2.1

This letter is to invite you to work with us to answer the question of whether screening for CrAg among PLHIV with severe immunodeficiency helps reduce mortality and improve retention in care.

With your participation, we hope the lessons learned will benefit practitioners in Vietnam and other countries in the region that are contemplating similar screening to provide the best care for their patients.

If you have any questions or want to know more, please contact Assoc. Prof Nguyen Van Kinh – National Hospital for Tropical Diseases or Dr Le Manh Hung – Tropical Diseases Hospital - Ho Chi Minh City representing the study team and VAAC.

| FOR | OPC |
|-----|--------------|
| | $\mathbf{O}$ |

### **APPENDIX 14A: SCREENING LOG FOR OPC**

| Clinic name: |
|--------------|
|--------------|

| No. | Participan<br>t name | OPC ID | Year<br>of<br>birth | Gender | Screening<br>date | Specimen<br>code | CD4 result<br>(cell /μL) | CrAg result | Be pregnant<br>/plan to be<br>pregnant | CrAg<br>released Date | Staff |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1. | | | | ☐ Male ☐ Female | | | | Positive Negative Not done | ☐ Yes<br>☐ No | | |
| 2. | | | | ☐ Male ☐ Female | | | | Positive Negative Not done | ☐ Yes<br>☐ No | | |
| 3. | | | | ☐ Male ☐ Female | | | | Positive Negative Not done | ☐ Yes<br>☐ No | | |
| 4. | | | | ☐ Male | | | | ☐ Positive ☐ Negative ☐ Not done | ☐ Yes<br>☐ No | | |
| 5. | | | | ☐ Male ☐ Female | | | | Positive Negative Not done | ☐ Yes<br>☐ No | | |
| 6. | | | | ☐ Male | | | | Positive Negative Not done | ☐ Yes<br>☐ No | | |
| 7. | | | | ☐ Male | | | | Positive Negative Not done | ☐ Yes<br>☐ No | | |

| CRICS study - #14E | Enrollment log | for OPC - | Ver 2.1 |
|--------------------|----------------|-----------|---------|
|--------------------|----------------|-----------|---------|

| <b>APPENDIX 14B:</b> | ENROLL | LMENT L | OG FOR | OPO |
|----------------------|--------|---------|--------|-----|
|----------------------|--------|---------|--------|-----|

| Clinic name: |
|--------------|
|--------------|

| No. | Participant<br>name | Year<br>of<br>birth | Gender | Phone<br>number of<br>participant | OPC<br>ID | CD4<br>result<br>(cell<br>/μL) | CrAg result | Agree to participate in the study | Enrollment<br>date | Study ID | Note |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | | | ☐ Male ☐ Female | | | | ☐ Positive ☐ Negative | ☐ Yes<br>☐ No | | | |
| 2 | | | ☐ Male ☐ Female | | | | ☐ Positive ☐ Negative | ☐ Yes<br>☐ No | | | |
| 3 | | | ☐ Male ☐ Female | | | | ☐ Positive ☐ Negative | ☐ Yes<br>☐ No | | | |
| 4 | | | ☐ Male ☐ Female | | | | ☐ Positive ☐ Negative | ☐ Yes<br>☐ No | | | |
| 5 | | | ☐ Male ☐ Female | | | | ☐ Positive ☐ Negative | ☐ Yes<br>☐ No | | | |
| 6 | | | ☐ Male ☐ Female | | | | ☐ Positive ☐ Negative | ☐ Yes<br>☐ No | | | |
| 7 | | | ☐ Male ☐ Female | | | | ☐ Positive | ☐ Yes<br>☐ No | | | |
| 8 | | | ☐ Male ☐ Female | | | | ☐ Positive ☐ Negative | ☐ Yes<br>☐ No | | | |

| Specimen code: |
|------------------------------------|
| OPC code: |
| YOB: Gender: |
| TEST DESIL T |
| TEST DESIL T |
| TECT DECLUT |
| TEST RESULT |
| Date month year 201 |
| Head of lab Department |
| Full name: |
| #15CrAg testing request form Ver 2 |
| STING FORM |
| Specimen code: |
| OPC code: |
| YOB: Gender: |
| TEST RESULT |
| Date month year 201 |
| Head of lab Department |

Full name:....

Full name:....

### **APPENDIX 16: CRAG TESTING LOG**

### FOR LABORATORY

### Laboratory name:

| No<br>· | Participant<br>name | Year<br>of<br>birth | Gender | Specimen<br>referral Unit | Specimen<br>receiving<br>date | Specimen code | CD4<br>result<br>(cell /μL) | CD4 indication | CrAg result | CrAg<br>released<br>Date | Screening conductor | Note |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1 | | | ☐ Male ☐ Female | | | | | ☐ New enrollment ☐ Routine monitoring ☐ Presumed treatment failure | Positive Negative Not done | | | |
| 2 | | | ☐ Male ☐ Female | | | | | New enrollment Routine monitoring Presumed treatment failure | Positive Negative Not done | | | |
| 3 | | | ☐ Male | | | | | ☐ New enrollment ☐ Routine monitoring ☐ Presumed treatment failure | Positive Negative Not done | | | |
| 4 | | | ☐ Male | | | | | New enrollment Routine monitoring Presumed treatment failure | Positive Negative Not done | | | |
| 5 | | | ☐ Male | | | | | ☐ New enrollment ☐ Routine monitoring ☐ Presumed treatment failure | Positive Negative Not done | | | |
| 6 | | | ☐ Male | | | | | New enrollment Routine monitoring Presumed treatment failure | Positive Negative Not done | | | |
| 7 | | | ☐ Male ☐ Female | | | | | New enrollment Routine monitoring Presumed treatment failure | Positive Negative Not done | | | |

### **APPENDIX 17: HEALTH-RELATED QUALITY OF LIFE FORM**

| Study ID | | | . 11 4 | Data | | | |
|---|---|---|---|---|---|---|---|
| | Add sticker | Date of | enrollment: | (full | name) | | |
| | here | /_ | | Signa<br>— | | | |
| Q | Quality of life | | | | | | |
| | TODA | AY | 1. Unable<br>to do | 2. Severe problems | 3. Moderate problems | 4. Slight problems | 5. No<br>problems |
| Q01 | Mobility | | | | | | |
| Q02 | Self-care | | | | | | |
| Q03 | Usual Activities study, housewo | ` • | | | | | |
| | leisure activitie | - | | | | | |
| | | | 1. Extremely | 2. Severely | 3.<br>Moderately | 4. Slightly | 5. None |
| Q04 | Pain / Discomf | fort | | | | | |
| Q05 | Anxiety / Depr | ression | | | | | |
| | We would like | Y. | | | | | |
| Q06 | This scale is no | umbered from 0 to 1 | 100. <b>100 means</b> | the best heal | th you can | | points |
| 200 | imagine; 0 me | eans the worst heal | th you can ima | igine. | | points | |
| | Please indicate | | | | | | |

### APPENDIX 18. PATIENT'S VISITS LOGBOOK

| Patient's ID: |
|---------------|
|---------------|

| | | | Number<br>of days<br>for which<br>ARVs<br>were<br>given | Any OIs since the last visit (using WHO clinical stages) | |
|---|---|---|---|---|---|
| Date of appointment | Actual date of visit | Medication<br>pick-up | | List all test-based<br>OIs diagnosed since<br>the last visit | List all clinical OIs diagnosed without any investigations since the last visit |
| // | _/_/ | ☐ Patient ☐ Family member | | | |
| // | _/_/ | ☐ Patient ☐ Family member | | | |
| // | _/_/ | Patient Family member | | | |
| // | _/_/ | Patient Family member | | | |
| // | _/_/ | Patient Family member | | | |
| // | _/_/ | ☐ Patient ☐ Family member | | | |
| // | _/_/ | Patient Family member | | | |
| _// | _/_/ | ☐ Patient ☐ Family member | | | |
| // | _/_/ | ☐ Patient ☐ Family member | | | |
| // | _/_/ | Patient Family member | | | |
| // | _/_/ | Patient Family member | | _ | _ |

### **APPENDIX 19. Fluconazole (pre-emptive treatment) log**

| Patient's | ID: | |
|-----------|-----|------|
| 1 aucht 3 | 110 | <br> |

| Phase | (Date of medication was given to | End date<br>(Date of<br>next<br>appointme<br>nt) | Dosage<br>(mg/day) | Formulation | Comments |
|---|---|---|---|---|---|
| Initial phase | | | | 150 mg x tablets ( tablets) 50 mg x tablets ( tablets) | |
| (2 weeks) | | | | 150 mg x tablets ( tablets) 50 mg x tablets ( tablets) | |
| | | | | ☐ 150 mg x tablets ( tablets) ☐ 50 mg x tablets ( tablets) | |
| Continuation phase | | | | 150 mg x tablets ( tablets) 50 mg x tablets ( tablets) | |
| (8 weeks) | | | | 150 mg x tablets ( tablets) 50 mg x tablets ( tablets) | |
| | | | | 150 mg x tablets ( tablets) 50 mg x tablets ( tablets) | |
| | | | | 150 mg x tablets ( tablets) 50 mg x tablets ( tablets) | |
| | | | | $ \begin{array}{ c c c c c c c c c c c c c c c c c c c$ | |
| | | | | $ \begin{array}{ c c c c c c c c c c c c c c c c c c c$ | |
| | | | | $ \begin{array}{ c c c c c c c c c c c c c c c c c c c$ | |
| Maintenance | | | | ☐ 150 mg x tablets ( tablets) ☐ 50 mg x tablets ( tablets) | |
| | | | | ☐ 150 mg x tablets ( tablets) ☐ 50 mg x tablets ( tablets) ☐ 150 mg x tablets ( tablets) | |
| | | | | 150 mg x tablets ( tablets) 50 mg x tablets ( tablets) | |
| | | | | $ \begin{array}{ c c c c c c c c c c c c c c c c c c c$ | |

### **CRICS study** - #19 Fluconazole (pre-emptive treatment) log - Ver 2.1

| End of therapy: Date/ |
|---|
| Reason to stop fluconazole(choose one item below): |
| $\square$ CD4 count $\ge$ 200 for more than 6 months |
| ☐ Viral load less than 1000 copies/mL(suppressed) in patient on ART for more than 6 months |
| Adverse drug reaction related to fluconazole |
| Other. Specify: |

### Appendix 20: Script informing patients of reimbursement

As you have agreed to join this study, we want to interview you about your feelings and some questions about your quality of life. Additionally, since you are spending some of your time with us for this interview, we'll reimburse you for this time. You will be reimbursed 65,000 Vietnam Dong for the extra time spent at the facility for study-related activities, including the time which is used to for answering the Quality of Life questionnaire. We pay you at the time of enrollment (baseline visit), and at 6 and 12 month), however you will not receive any reimbursement for your previous visits to OPC.

### **APPENDIX 21: COST STUDY DATA COLLECTION TOOLS**

See Excel files enclosed